CLINICAL TRIAL: NCT00919373
Title: Substrate Modification in Stable Ventricular Tachycardia in Addition to ICD Therapy
Brief Title: Substrate Modification in Stable Ventricular Tachycardia in Addition to Implantable Cardioverter Defibrillator (ICD) Therapy
Acronym: VTACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T46
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Ventricular Tachycardia; Coronary Artery Disease; Left Ventricular Dysfunction
Keywords: Catheter Ablation; Defibrillators, Implantable
MeSH Terms: conditions — Tachycardia, Ventricular; Coronary Artery Disease; Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICD-Implantation (Active Comparator): Implantation of an Implantable Cardioverter Defibrillator (ICD) alone.
  Interventions: Procedure: ICD Implantation
- ICD + Ablation (Active Comparator): Stratified Catheter Ablation of Ventricular Tachycardia and ICD Implantation
  Interventions: Procedure: Substrate modification; Procedure: VT ablation; Procedure: ICD Implantation

INTERVENTIONS:
Procedure: Substrate modification — Catheter Ablation procedure - Substrate modification in sinus rhythm in case of unstable induced monomorphic Ventricular Tachycardia (VT) which does not allow mapping and ablation in tachycardia, or noninducible stable clinical VT.
  Arms: ICD + Ablation
Procedure: VT ablation — Catheter Ablation of Ventricular Tachycardia (VT) in case of stable VT
  Arms: ICD + Ablation
Procedure: ICD Implantation — Implantation of a marked released Implantable Cardioverter Defibrillator manufactured by St. Jude Medical

SUMMARY:
The main objective of this study is to compare the time from randomization to the first recurrence of any ventricular tachycardia (VT) in patients undergoing VT ablation (for stable VTs) and substrate ablation (for unstable VTs) after an initial episode of stable VT and patients not undergoing ablation, with both groups under the protection of an ICD.

DETAILED DESCRIPTION:
The main objective of this study is to compare the time from randomization to the first recurrence of any VT in patients undergoing VT ablation (for stable VTs) and substrate ablation (for unstable VTs) after an initial episode of stable VT and patients not undergoing ablation, with both groups under the protection of an ICD.

Prior to the ablation, the patients will undergo electrophysiologic study (EPS) with programmed ventricular stimulation, with the aim to reproduce the clinical VT. Most patients with coronary artery disease, systolic LV dysfunction, and one episode of clinical sustained VT have more than one inducible VT at electrophysiologic study. Since any inducible VT can become a potential clinical VT (24), an attempt will be made to ablate the clinical stable VT, as well as all inducible morphologies, stable or unstable.

One of the following 2 ablation strategies will be possible for each VT:

* Substrate modification in sinus rhythm in case of unstable induced monomorphic VT which does not allow mapping and ablation in tachycardia, or noninducible stable clinical VT.
* VT ablation in tachycardia in case of stable VT

For each procedure the number of tachycardias , the type of each tachycardia (inducible or noninducible, stable or unstable), the ablation strategy for each tachycardia (it is possible that lesions deployed for one tachycardia will render another tachycardia noninducible as well) and the procedural outcome for each tachycardia will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease For the purpose of this study, coronary artery disease will be defined as the presence of a 50 % or more diameter stenosis of the left main coronary artery, or 75 % or more diameter stenosis of the left anterior descending, circumflex or right coronary arteries, or the history of a surgical or percutaneous revascularization procedure, or history of successful thrombolysis, or a history of prior myocardial infarction (e.g.: documented by Q-wave, R-reduction, aneurysm)
* Left ventricular ejection fraction ≤ 50 % as estimated by echocardiography or contrast ventriculography within the previous 30 days and evidence for old myocardial infarction (ECG, echocardiographic or venticulographic).
* One episode of documented stable clinical VT without any reversible causes
* Written informed consent

Exclusion Criteria:

* Age < 18 years or > 80 year
* Protruding LV thrombus on pre-ablation echocardiogram
* Acute myocardial infarction within the preceding 1 months
* Class IV NYHA heart failure
* Valvular heart disease or mechanical heart valve precluding access to the left ventricle
* Unstable angina
* Cardiac surgery involving cardiotomy (not CABG) within the past 2 months
* Serum creatinine > 220 mmol/L (2.5 mg/dL)
* Thrombocytopenia or coagulopathy
* Contraindication to heparin
* Pregnancy
* Acute illness or active systemic infection
* Other disease process likely to limit survival to less than 12 months
* Significant medical problem that in the opinion of the principal investigator would preclude enrollment in the study
* Participation in another investigational study
* Unwillingness to participate or lack of availability for follow-up
* Incessant VT or electrical storm
* Bundle branch reentry tachycardia as the presenting VT
* Preexisting ICD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2002-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
recurrence of any sustained clinical VT, stable or unstable, monomorphic or polymorphic, including VF, during the follow-up period | 2 years

SECONDARY OUTCOMES:
Severe clinical events (death, number of syncopes, number of hospital admissions for a cardiac indication, number of episodes of electrical storm (more than 3 VT episodes in 24 hours)) during the follow-up period . | 2 years
Quality of life | 2 years
Number of adequate ICD interventions (shocks and overdrive episodes caused by recurrence of VT or VF and not supraventricular arrhythmias or mechanical lead problems). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, Prof. Dr., Principal Investigator — Asklepios Klinik St. Georg, Hamburg, Germany
Locations (16):
- Institute for Clinical and Experimental Medicine, Prague, Czechia
- University Hospital of Aarhus, Aarhus, Denmark
- Germany (13):
  - Universitäts Medizin Mannheim, Mannheim, Baden-Wurttemberg
  - Herz- und Gefäßklinik Bad Neustadt, Bad Neustadt an der Saale, Bavaria
  - Klinikum Großhadern der Ludwig-Maximilians-Universität München, München, Bavaria
  - Kerckhoff Klinik GmbH, Bad Nauheim, Hesse
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Medizinische Einrichtungen der Rheinischen Friedrich-Wilhelm-Universität, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Helios Klinikum Wuppertal Klinikum Barmen, Wuppertal, North Rhine-Westphalia
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Medizinische Fakultät der Universität Magdeburg, Magdeburg, Saxony-Anhalt
  - Asklepios Klinik St. Georg, Hamburg
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Klinikum der Ruprecht-Karls-Universität Heidelberg, Heidelberg
- Universitätsspital Bern, Bern, Switzerland

REFERENCES:
- [Result] Kuck KH, Schaumann A, Eckardt L, Willems S, Ventura R, Delacretaz E, Pitschner HF, Kautzner J, Schumacher B, Hansen PS; VTACH study group. Catheter ablation of stable ventricular tachycardia before defibrillator implantation in patients with coronary heart disease (VTACH): a multicentre randomised controlled trial. Lancet. 2010 Jan 2;375(9708):31-40. doi: 10.1016/S0140-6736(09)61755-4. PMID 20109864